CLINICAL TRIAL: NCT01667328
Title: Utility of Preoperative Massage in Breast Surgery Patients
Brief Title: Preoperative Massage in Breast Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vassar Brothers Medical Center (Other)
Collaborators: Health Quest Systems (Unknown); Dyson Center for Cancer Care (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012-2
Record Dates: First submitted 2012-06-14; First posted 2012-08-17 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Anxiety; Presurgical Anxiety; Breast Cancer
Keywords: Anxiety; Presurgical anxiety; Breast Cancer
MeSH Terms: conditions — Anxiety Disorders; Breast Neoplasms | interventions — Massage; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Massage therapy (Experimental): This group will received presurgical massage
  Interventions: Procedure: Massage therapy
- Control (Placebo Comparator): Standard of care with no massage
  Interventions: Procedure: Standard of care

INTERVENTIONS:
Procedure: Massage therapy — Presurgical 15 minute massage performed by a licensed massage therapist
  Arms: Massage therapy
Procedure: Standard of care — Control group will receive standard of care with no massage therapy
  Arms: Control

SUMMARY:
This randomized controlled interventional study is designed to determine whether breast cancer surgical patients receiving presurgical massage therapy performed by a licensed massage therapist have decreased average anxiety levels compared to the control group of breast cancer surgical patients who do not receive massage therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Must speak English
* Able to give consent
* 18 years of age or older
* Undergoing first procedure outpatient breast/axillary surgery at Vassar Brothers Medical Center

Exclusion Criteria:

* Anxiolytics or antidepressants medications during the previous 24 hours
* Any condition that would prohibit receiving a massage
* IV medications prior to presurgical holding VAS assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2012-06; Primary Completion 2018-03 (Actual); Study Completion 2018-03-19 (Actual)

PRIMARY OUTCOMES:
Anxiety level | Upon arrival at the hospital for scheduled surgery and again immediately prior to surgery. Expected interval between measurements estimated to be less than 120 minutes.
  Assessments will be done immediately post registration and immediately prior to surgery

CONTACTS AND LOCATIONS:
Overall Officials: Angela Keleher, M.D., Principal Investigator — Vassar Brothers Medical Center
Locations (1):
- Vassar Brothers Medical Center, Poughkeepsie, New York, United States